CLINICAL TRIAL: NCT05935813
Title: Characteristics of Adolescents Affected by Dental Caries
Brief Title: Caries in Adolescents (Karies Hos Ungdom)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kompetansesenteret Tannhelse Midt (TkMidt) (Other)
Collaborators: Norwegian University of Science and Technology (Other); SINTEF Health Research (Other); Trøndelag Fylkeskommune (Unknown); University of Sheffield (Other); Karolinska Institutet (Other); Ablemagic AS (Unknown); Orkla Care AB (Industry); UiT The Arctic University of Norway (Other); University of Bergen (Other); Forandringsfabrikken (Unknown)
Responsible Party: Sponsor
Other Study IDs: 217487 Karies hos ungdom
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Caries,Dental
Keywords: Caries; Adolescents; Caries risk factors
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- 1996 birth year: Followed cohort for 6 years (2008-2014) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries
- 1997 birth year: Followed cohort for 6 years (2009-2015) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries
- 1998 birth year: Followed cohort for 6 years (2010-2016) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries
- 1999 birth year: Followed cohort for 6 years (2011-2017) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries
- 2000 birth year: Followed cohort for 6 years (2012-2018) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries
- 2001 birth year: Followed cohort for 6 years (2013-2019) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries
- 2002 birth year: Followed cohort for 6 years (2014-2020) to study time trends in caries experience
  Interventions: Other: Study characteristics of adolescents affected by dental caries

INTERVENTIONS:
Other: Study characteristics of adolescents affected by dental caries — Study and compare data from The Trøndelag Health Study (The HUNT Study) and data from Public dental service records in Trøndelag collected 2008-2020 to look for Characteristics of adolescents affected by dental caries and trends in caries experience among adolescents (12-20 yo).

SUMMARY:
In this study the objective is to establish in depth knowledge about adolescents' oral health characteristics, - practices and - needs. Further, we want to evaluate whether adolescents' caries status can be associated with existing socio-economic inequality, emotional health and lifestyle factors.

The main question[s] it aims to answer are:

1. What is the caries status (i.e. prevalence, increment at different timepoints and characteristics) among adolescents in Trøndelag?

   * What is the caries prevalence in different age groups?
   * Is there any difference in caries prevalence linked to specific age groups, gender or urban versus rural areas?
   * Are approximal tooth surfaces especially prone to the development of new caries lesions?
   * Is the caries increment from 12 to 20 years a continuous process or are there high-risk periods within this timespan?
   * How is the prevalence of enamel caries? Is enamel caries more prevalent in younger age groups than in older age groups?
2. What are the patterns of recall intervals and non-attendance in different age groups, among adolescents in Trøndelag?

   * What are the attendance rates and prevalence of non-attendance at dental appointments in different age groups?
   * What is the recall interval between regular follow-up dental visits?
   * Are there any recall or attendance characteristics linked to age group, gender or urban versus rural areas?
3. What factors (i.e. oral health behaviours, socioeconomic-, lifestyle- and parental factors) are associated with caries among Norwegian adolescents?

   * How are the oral health behaviours (i.e. dietary- and oral hygiene habits, attendance to dental care) among adolescents, and are there any shared oral health behavioural challenges?
   * Is the caries prevalence linked to life challenges (mental illness, alcohol/drug use and chronic diseases)?
   * To what degree are oral health behaviours associated with caries among adolescents?
   * Is there any association between media screen time and oral health behaviours, and cariesstatus?
   * Is there any association between physical activity, sport participation and oral health behaviours, and caries status?
   * What are the associations between socioeconomic factors (study program, birth- and migration background, and parental income, education and employment) and oral health behaviours, and caries status?

For research question 1 and 2, the sample will be adolescents aged 12-20 years living in Trøndelag county in the time period 2008-2020, (n≈115000, Statistics Norway, SSB). Data will be extracted from dental health records in the public dental service (Den offentlige tannhelsetjenesten, Trøndelag Fylkeskommune).

The public dental service annually reports caries prevalence for 12- and 18-year-olds, Statistics Norway, SSB (Figure 1). However, the knowledge is modest about the caries development within the six years from 12 to 18 years of age. Further, the public dental service offers subsidised dental care to 19- and 20-year-olds. Extracting data from dental health records in the public dental service will give us the opportunity to explore the caries increment at multiple timepoints, and attendance rates at dental appointments throughout the teenage period from 12 to 20 years of age.

For research question 3, the sample will be adolescents (n≈8000) and their parents that participated in the fourth survey of The Trøndelag Health Study (HUNT4) in 2017-2019. Self-reported questionnaire data will be linked to data from dental health records in the public dental service.

DETAILED DESCRIPTION:
Characteristics of adolescents affected by dental caries Substudy of #Care4YoungTeeth<3 Relevance A modern definition of oral health includes, in addition to disease and condition status, underlying determinants, moderating factors, overall health and well-being. This means that the definition also encompasses the ability to speak, smile, smell, taste, touch, chew, swallow and express emotions,and functioning without feeling pain or discomfort.

In this study dental caries will be targeted, being widespread in the teenage population. In Northern Norway a recent publication among 16-year-olds concluded that caries (enamel caries included) constituted a major health problem and affected the total teenage population. This means that adolescence is a vulnerable period concerning initiation and progression of caries. As it is known, when caries are initiated but still has not reached dentin layer, restorations can be avoided. Seen in light of life-perspective, to target adolescence, is essential when the objective is to improve oral health into adulthood and reduce repair costs for re-doing restorations.

Caries into dentin layer is skewed distributed i.e. individuals living in vulnerable populations as in families with low income, in some immigrant minorities and where these two populations overlap, are those carrying the majority of caries burden. These groups also appears to have less benefit from universal promotive- and preventive strategies when compared to the general population.Therefore, these adolescents need both a general population-based and simultaneously an additional high-risk prevention approach. A challenge is to identify these groups, but authors have identified groups at caries risk successfully by linking caries data to socio-cultural- and socio-economic official data or to use geographic maps ("Geo-map").

Adolescence is described as a period of continued behavioral development along a pathway established in childhood, and during this period the behavior patterns differ from both childhood and adulthood. Characteristics of the period are peer interactions, frequent conflicts and opposition towards either parents, teachers or both, as well as increased risk-taking behaviors, depression and anxiety. According to Statistics Norway 2019, among the group children and adolescents living in Norway, 759 68 are immigrants and 133 315 are of immigrant origin (born in Norway, but with immigrant parents). There are reasons to believe that adolescents living in cultural minorities have a daily life different from their peers in the general population, both in respect to food/drinking habits, frequency of meals and other oral health habits influenced by culture. Time trends not only influence an oral disease alone, but also the determinants behind the disease.How do the oral diseases appear during recent years? Do any time trends appear when comparing nowadays disease status with previous corresponding data? Are during recent years background oral disease determinants changed? Which characteristics represent the high-risk individuals? Background and status of knowledge Dental Caries National oral health data reported in Norway and Sweden are limited to caries at dentin level, a system which underscores the true caries experience. However, these data give us valuable information and enable comparisons between the two neighboring countries. In 2019, 19% of Norwegian 5-year-olds, 36% of 12-year-olds and 71% of 18-year-olds experienced caries at dentin level. Geographic variations were substantial; the highest proportion of 18-year-olds (83%) from previous Finnmark county and the lowest (65%) from previous Hedmark county. Comparing 2019 statistics of young individuals with a previously evaluation of corresponding caries data up to 2005, it seems that the overall trend of caries reduction during recent years mainly has taken place before the age of 12 years. The proportion of 18-year-old with caries at dentin level in previous Finnmark county in 2019, is almost identical to the corresponding proportion registered in 2005. This means that adolescence is a caries preventive resistant period. It is worth to be mentioned that this reduction seen before 12 years of age, may in part be due to the trend change in diagnostic and treatment caries criteria which today is more conservative than before.

There are some explicable reasons why first part of adolescence is a risk period for caries. At 12 years of age, many teeth have just emerged and thus due to immature outer enamel, categorized as a caries prone age. Individuals of 12-15 years are also shown to develop more new enamel lesions on approximal surfaces when compared to young adults. The permanent second molar has its highest risk period during the first 3 years after the eruption (12-15 years). Additionally, distribution of caries (at dentin level) at approximal surfaces has shown skewness with some surfaces more caries prone than others, especially distal surface of the second permanent premolar.

However, this meticulous work was done more than twenty years ago, which means that it is not sure the findings reflect the caries tooth surface distribution of today. A Norwegian study has also documented the second premolars to be responsible for the majority of caries increment at dentin level from the age 12 to 18 years. National data from Sweden showed caries approximal surfaces to affect 31% of 19-year-olds (Socialstyrelsen), but when including enamel carries as done in a Swedish study, a different picture emerged. This study presented approximal initial caries in 15- year-olds to be 6 times more prevalent than manifest lesions and fillings, constituting 86% of the total number of approximal caries lesions. This finding is important, emphasizing the potential of preventive dental strategies among adolescents. Updated knowledge of which surfaces are most prone to caries, and at a stage of caries development before the dentin layer, should be highly prioritized.The rate of the lesion progression is expressed as the survival time. In a low caries prevalence population, it takes 3 years (median survival time) before a lesion at the enamel-dentin border progress into the dentin. Only half of these lesions progressed into dentin during this time, while the other half did not. When we also include the time period for caries initiation at a surface and the time period for progression into the enamel-dentin border, there is sufficient time to interact before dentin layer is reached. It is therefore important already from early adolescence to prioritize promotion and prevention. If lesions can be prevented from reaching into dentin in adolescence, the risk of progression into dentin significantly diminishes after 20 years of age. However, caries progression increases when the caries prevalence is high, so for high risk adolescents, the time period to reach the dentine layer is shorter compared to their peers in the general population. We also know, if the prevalence at dentin level is high, dentin lesions according to Nigel Pitts, represent only the top of a "caries iceberg", of which enamel caries constitutes the wide baseline. One method to identify individuals with high caries experience, is to use the Sic-index reported at the age of 12 years (the Mean DMFT of the one third of the study group with the highest caries score). Oral health risk assessment It is of most importance to identify caries determinants/risk factors and potential interactions between them, both for the general adolescent population and for those at high risk. Adolescence is considered to be the period in which many behaviors and attitudes are molded, included those of oral health. If we do not know which background factors are present, both promotion and prevention will fail because the social circumstances of the individual or family is a barrier forbehaviour change. Determinants are additive; the more determinants present, the higher risk for disease development. Socioeconomic background The society is changing and with it, its populations and their oral health determinants. As the adolescents' behaviour is based on a pathway established in childhood, the current style of parenting and pattern of family life when compared with previous decades, also have changed and today represent other oral health determinants than before. "Democratic up-bringing" as being allowed to negotiate about what and when to eat, parental indulgence etc. are more frequent than before. Low socio-economic background, however, has for years been shown to be associated with unfavorable oral health and still contributes a potent oral health determinant, even in countries with free dental care. Socio-economic inequalities, though more visible in younger age groups, are present also among adolescents. Subgroups with extra life challenges A trait of today is that many adolescents drop high school without having a job to go to, which negatively affects their self-esteem. Society targets on success in all ways, make many teenagers depressed or give them feelings of not fitting in or being excluded from society. Especially among teenage girls, it is debated whether mental illness is increasing or not. Norwegian Institute of Public Health in 2018 reported that during the period 2008-2011 around 5% of 15-17-year-girls had a diagnosis of mental illness while the corresponding prevalence had increased to 7% in 2016. A side-effect of psychoactive drugs is xerostomia, which means reduced saliva protection against both caries. Other mental health conditions, e.g. eating disorders are not uncommon, especially among girls. A study including participants from 15 years of age, found eating disorders especially high in female athletes and in leanness-dependent sports. In respect to these disorders, connected behaviours and diet are found harmful for oral health, for erosion in particular.Use of illegal narcotics and dependency also are problems during adolescence, and teenagers affected can after short period experience teeth destruction. In 2019, the National Institute of Public Health, Norway, reported that 26.4% of the age group 16-24 years, had used cannabis at least once, while in case of amphetamine and of ecstasy/MDMA, the percentages were 1.4% and 3.7%, respectively. Oral health behaviour - dietary habits From 13 years up to 19 years, differences in lifestyle, maturity and priorities are observed. The older, the more they make their own decisions influenced by their own priorities and not so much as before prone to parental influence. Many also in the end of adolescence leave home to live alone. In society of today, fast food and soft-drinks are easily accessible and irregular meals have become a trend of modern lifestyle. Many adolescents due to this lifestyle, suffer from overweight and obesity, both conditions linked to caries development. Beverage related sugar intake are documented to be related to electronic device use, constituting threats for initiating caries.

Oral health behaviour - oral hygiene habits During adolescence peers and neighbourhood increase their influence, so the environment they happen to socialize within, might affect their oral behavioural habits, e.g. oral hygiene behaviours. In a study among 14-year-olds recently published, most teenagers did not daily use dental floss, fewer boys than girls. Among students in secondary education (8-13 years of school) in western Norway in 2016, 65.2% of those of 11-13 grade reported that they brushed their teeth more than once a day, and boys showed a significantly lower percentage than girls. In a study among Swedish 19-year-olds, also boys were significantly less likely to not perform daily tooth-brushingtwice or more than girls. Out of the same 19-year-olds, those with high scores of plaque and gingivitis, also had a less positive perceptions, attitude and behaviours towards oral health than those with favourable oral hygiene conditions. Oral health behaviour - non-attendance to dental care Non-attendance to dental care are more frequent among boys and by older children. One Norwegian study suggested that reasons could be that older adolescents make their own priorities and can have difficulties to leave studies and jobs for dental visits. Dental anxiety has also been reported to be associated with non-attendance to dental care. In Swedish Specialized Paediatric Dentistry non-attendance has also been observed among adolescents with dental behavioural management problems (DBMP). Furthermore, negative attitudes towards dental personnel is reported to contribute to dental avoidance. A constructed variable "Few missed dental appointments" has among Swedish 19-year-olds found to positively associated with daily tooth-brushing twice or more. Missed dental appointments and non-regular dental care have also by many researchers been connected with poorer oral health or emergency care among children.

This means that during the adolescence period, a focus is needed on socioeconomic background, subgroups with extra life challenges, various oral health behaviour as dietary- and oral hygiene habits, and non-attendance to dental care. To improve some existing oral health behaviours as oral hygiene routines, especially boys should be targeted. We also have to acknowledge that subgroups of adolescents are struggling in various ways, negatively impacting their oral health. As oral health workers, we must see these adolescents as subjects and be informed about what their oral health challenges are. Otherwise, we cannot adapt our health care messages.#Care4YoungTeeth<3 The study described in the current protocol is a substudy of a larger research project,

* Care4YoungTeeth<3 (supplementary file, NRC project proposal), aiming to establish tailored oral health preventive strategies for adolescents at oral health high risk, and to establish universal oral health strategies for the adolescent group as a whole. The project management of
* Care4YoungTeeth<3 is based at SINTEF. This application concerns the first work package in
* Care4YoungTeeth<3 (WP1, task 1.1, described in brief in the NRC proposal, page 5), in which TkMidt is the responsible partner. Separate REC approval applications for subsequent work packages will be submitted later. Objectives In this study the objective is to establish in depth knowledge about adolescents' oral health characteristics, - practices and - needs. Further, we want to evaluate whether adolescents' caries status can be associated with existing socio-economic inequality, emotional health and lifestyle factors. The results from this study will guide the further process of co-creating new products, tools, and service touchpoints in the main project, #Care4YoungTeeth<3.The HUNT Study The Trøndelag Health Study (The HUNT Study) is a large population-based cohort study conducted in Norway. The HUNT Study has been repeated about every ten years; HUNT1 1984-86, HUNT2 1995- 97, HUNT3 2006-08 and HUNT4 2017-19. Adolescents were included in the second HUNT survey, in 1995-97. A follow-up was arranged in 1999-2000, The Young-HUNT2 Survey. In 2006-2008 The Young-HUNT Survey was again an integrated part of The HUNT Study, this time the third HUNT survey and the third Young-HUNT survey (44). The Young-HUNT4 Survey, 13-19-year-olds, was performed at schools in the region. Participants not attending school were invited to join the survey at the field station in their municipality. Hence, all residences, 13 years and older, in then Nord-Trøndelag county were invited to participate in HUNT4. The county is mostly rural, with no large cities, but is in many ways representative of Norway regarding geography, economy, industry, and sources of income, age distribution, morbidity and mortality. Every participant is thoroughly mapped with regards to physical health, mental health and lifestyle, building a unique database of questionnaire data, clinical measurements and samples from the county's inhabitants from 1984 onwards, the HUNT databank (https://hunt-db.medisin.ntnu.no/hunt-db/#/). Dental health records Oral health data will be extracted from dental health records in the public dental service (Den offentlige tannhelsetjenesten, Trøndelag Fylkeskommune). We will use clinical measures of dental status (DMFT/S) (both when enamel caries is included and not), as well as information on the use of dental services such as frequency of appointments and missed appointments. Statistical analysis Simple descriptive statistics of frequencies and proportions will be used to assess dental caries status in different age groups. To inspect univariate differences, chi-square tests (for categorical variables) or independent t-tests (for continuous variables) will be used. To assess the impact of various factors on dental caries experience, adjusting for confounders, the negative binomial hurdle model will be applied. The hurdle model is one of the recommended models for outcome distributions with an excessive number of zeros, like is typically the case when studying caries as an outcome. The hurdle models consists of both a logistic regression part that assesses the prevalence of the outcome according to the exposure (like whether a child experiences caries or not), and a negative binomial distribution that assesses the degree of caries experience for those with caries experience. To assess the incidence of new caries, survival analyses by Cox Regression and Kaplan-Meier curves will be performed, given that the proportionality assumption is satisfied, otherwise other appropriate methods will be used. The analyses will be performed using statistical software (SPSS, STATA or R).

Project organization and management The current project is one of the tasks in the first work package in #Care4YoungTeeth<3. Center for Oral Health Services and Research (Kompetansesenteret Tannhelse Midt, TkMidt) is the responsible partner for this task and will provide dental and epidemiological expertise. Project members (Tone Natland Fagerhaug, PhD, senior researcher; Hedda Høvik, PhD, dentist/researcher; Marit Slåttelid Skeie, dentist/professor emeritus; Ingrid Berg Johnsen, psychologist/PhD-candidate, Abhijit Sen epidemiologist/reseacher). Collaborating partners: SINTEF AS (Marikken Høiseth, PhD, researcher/designer, project manager; Anita Das, PhD, research manager; Kristine Holbø, MSc, senior researcher/designer; Eva Lassemo, PhD, researcher; Kari Sand, PhD, senior researcher), Trøndelag county (Bjørnar Hafell, assistant county director for Dental Health), University of Tromsø (Jan-Are K.

Johnsen, associate professor.), University of Sheffield (Zoe Marshman, professor; Helen Rodd, professor), Karolinska Institutet (Göran Dahllöf, dentist/professor). The research group is a multidisciplinary collaboration including comprehensive competency in fields like oral health research, paediatric dentistry and epidemiology.Publications: tentative titles

1. Caries incidence at different timepoints during adolescence from age 12 in Trøndelag.
2. Patterns of dental appointment intervals and non-attendance from age 12 to 20 years in Trøndelag.
3. Background caries determinants and oral health behaviours in adolescents - The Young HUNT4 study.
4. Caries prevalence in adolescents with various life challenges - to what extent do these challenges impact on caries prevalence? The Young HUNT4 study. Budget The funding needed for this work package is mainly associated with wages for those who will be employed in the project. For the employees at TkMidt, the costs will be funded through the Norwegian Directory of Health's funding scheme for the public regional oral health centers in Norway. Trøndelag county, University of Tromsø, University of Sheffield and Karolinska Institutet will cover their own expenses. SINTEF has applied for funding for the project #Care4YoungTeeth<3 (all work packages) through the Norwegian Research Council call KSP20PD. We expect there to be a high probability that the project will be funded, as oral health is one of the highlighted topics in this call. However, the work package described here will be conducted regardless of other external funding is granted or not.Ethics For research question 1 and 2, the ethical question comes to privacy considerations as we want to use information stored in the patient's dental records for research without consent. We seek exemption from the duty of confidentiality (Health Research Act § 35) for the extraction of dental health data from patient records, due to the large number of participants (n>150000) making obtaining consent difficult. Nevertheless, we believe that the participants' welfare and integrity is safeguarded. The data will be extracted in anonymous form and will thus emerge as anonymous information for the researchers. The information is equivalent the information already reported to the annual KOSTRA statistics/KPR registry, but with the difference that we also wish to include information on age, gender and municipality. Caries data and dental appointment attendance information collected for the current study, are not considered to be particularly sensitive.

Information about caries status and attendance rate for selected age groups (5, 12, and 18 years old) at the county level is annually reported to KOSTRA/KPR registry due to its public health importance.

We wish to include all the age groups between 12 and 20 years, in order to study whether there are critical timepoints during the adolescence for caries development. Such findings will form important background data when establishing future caries preventive strategies and interventions. Given that caries is one of our public health concerns, it could be argued that the benefits of the study outweigh the disadvantages related to extracting data from dental records without obtaining the participants consent. For research question 3, we will use data from Young-HUNT, linked to HUNT-data from their dental health records and their parents. Participants in The HUNT Study have signed a written consent regarding the screening and the use of data for research purposes, including the use of data fromdental health records. The HUNT4 data collection was approved by the Norwegian Data Inspectorate.

This research project will seek approval from the Regional Committees for Medical and Health Research Ethics (REK). This project will only use data from surveys and examinations that has already been performed.

Hence, the participants will not be exposed to additional screenings. Results from the study will be presented at group level. We will ensure that the analysis is performed thoroughly and that the results are published with care, without violating the integrity of individuals or groups.

As researchers, we find that it is an ethical obligation to use the data collected in The HUNT Study to gain more knowledge about dental status and possible oral health risk factors among adolescents in Norway. Here, especially to guide the enhancement of oral health preventive strategies for adolescents in #Care4YoungTeeth<3. Data management HUNT Databank generates a pseudo anonymized dataset based on the variables needed in the project. The dataset from HUNT Databank and the analysis generated in the project will be stored under access restriction on servers in the IT system at TkMidt. The IT services at TkMidt are responsible for daily back-ups of servers. Documentation on the analysis performed will be retained for a period of five years after the final study report/publication, unless otherwise decided by REK. Following final publications, the data will be stored under access restriction on servers in the IT system at TkMidt. All data is pseudo anonymized, and the identification key will be stored at a different institution, HUNT Databank.

ELIGIBILITY:
Inclusion Criteria:

* Patients born 1996-2002 registered in Public dental service(PDS) in the Trøndelag county. Adolescents aged 12-20 years living in Trøndelag county in the time period 2008-2020,

Exclusion Criteria:

* Adolescents aged 12-20 years living in Trøndelag county in the time period 2008-2020, not registered in PDS in this time period

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Adolescents aged 12-20 years living in Trøndelag county in the time period 2008-2020,
Sampling Method: Probability Sample
Enrollment: 115000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
Caries increment at dentine level | Six years
  Difference in caries experience at dentine level from 12 to 18 years of age
Enamel caries increment | Six years
  Difference in enamel caries increment from 12 to 18 years of age

SECONDARY OUTCOMES:
Baseline caries experience - impact on increment | six years
  Does baseline caries experience at 12 years impact increment?
Impact on increment - sex | six years
  Does sex impact increment?

CONTACTS AND LOCATIONS:
Locations (1):
- TkMidt, Trondheim, Trøndelag, Norway

REFERENCES:
- [Background] Glick M, Williams DM, Kleinman DV, Vujicic M, Watt RG, Weyant RJ. A new definition for oral health developed by the FDI World Dental Federation opens the door to a universal definition of oral health. J Am Dent Assoc. 2016 Dec;147(12):915-917. doi: 10.1016/j.adaj.2016.10.001. No abstract available. PMID 27886668
- [Background] Jacobsen ID, Crossner CG, Eriksen HM, Espelid I, Ullbro C. Need of non-operative caries treatment in 16-year-olds from Northern Norway. Eur Arch Paediatr Dent. 2019 Apr;20(2):73-78. doi: 10.1007/s40368-018-0387-z. Epub 2018 Dec 4. PMID 30515661
- [Background] Raadal M, Espelid I, Crossner C. Non-operativ vs operativ behandling av karies blant barn og unge. Er det tid for å endre strategi? Den Norske Tannlegeforeningens Tidende. 2011;121:10-7.
- [Background] Isaksson H, Alm A, Koch G, Birkhed D, Wendt LK. Caries prevalence in Swedish 20-year-olds in relation to their previous caries experience. Caries Res. 2013;47(3):234-42. doi: 10.1159/000346131. Epub 2013 Jan 11. PMID 23328627
- [Background] Socialstyrelsen S. Sociala skillnader i tändhälsa blnd barn och unga. Underlagsrapport till Barns och ungas hälsa, vård och omsorg. 2013. 2013.
- [Background] Skeie MS, Klock KS. Dental caries prevention strategies among children and adolescents with immigrant - or low socioeconomic backgrounds- do they work? A systematic review. BMC Oral Health. 2018 Feb 7;18(1):20. doi: 10.1186/s12903-018-0478-6. PMID 29415706
- [Background] Christensen LB, Twetman S, Sundby A. Oral health in children and adolescents with different socio-cultural and socio-economic backgrounds. Acta Odontol Scand. 2010 Jan;68(1):34-42. doi: 10.3109/00016350903301712. PMID 19878044
- [Background] Stromberg U, Magnusson K, Holmen A, Twetman S. Geo-mapping of caries risk in children and adolescents - a novel approach for allocation of preventive care. BMC Oral Health. 2011 Sep 26;11:26. doi: 10.1186/1472-6831-11-26. PMID 21943023
- [Background] Novak A, Pelaez M. What is adolescent behavioral development? In: Novak A, Pelaez M, editors. Child and adolescent development A behavioral systems approach. London: Sage Publications, Inc.; 2004. p. 463-92
- [Background] Skeie MS, Klock KS. Scandinavian systems monitoring the oral health in children and adolescents; an evaluation of their quality and utility in the light of modern perspectives of caries management. BMC Oral Health. 2014 Apr 30;14:43. doi: 10.1186/1472-6831-14-43. PMID 24885243
- [Background] Haugejorden O, Birkeland M. Karies i Norge i fortid og fremtid: Analyse av endringer og årsaker. Nor Tannlegeforen Tid. 2008;118:84-90
- [Background] Vidnes-Kopperud S, Tveit AB, Espelid I. Changes in the treatment concept for approximal caries from 1983 to 2009 in Norway. Caries Res. 2011;45(2):113-20. doi: 10.1159/000324810. Epub 2011 Mar 17. PMID 21412003
- [Background] Mejare I, Kallest l C, Stenlund H. Incidence and progression of approximal caries from 11 to 22 years of age in Sweden: A prospective radiographic study. Caries Res. 1999;33(2):93-100. doi: 10.1159/000016502. PMID 9892776
- [Background] Mejare I, Stenlund H, Zelezny-Holmlund C. Caries incidence and lesion progression from adolescence to young adulthood: a prospective 15-year cohort study in Sweden. Caries Res. 2004 Mar-Apr;38(2):130-41. doi: 10.1159/000075937. PMID 14767170
- [Background] Mejare I, Kallestal C, Stenlund H, Johansson H. Caries development from 11 to 22 years of age: a prospective radiographic study. Prevalence and distribution. Caries Res. 1998;32(1):10-6. doi: 10.1159/000016424. PMID 9438566
- [Background] David J, Raadal M, Wang NJ, Strand GV. Caries increment and prediction from 12 to 18 years of age: a follow-up study. Eur Arch Paediatr Dent. 2006 Mar;7(1):31-7. doi: 10.1007/BF03320812. PMID 17140525
- [Background] Alm A, Wendt LK, Koch G, Birkhed D. Prevalence of approximal caries in posterior teeth in 15-year-old Swedish teenagers in relation to their caries experience at 3 years of age. Caries Res. 2007;41(5):392-8. doi: 10.1159/000104798. PMID 17713340
- [Background] Pitts NB. Are we ready to move from operative to non-operative/preventive treatment of dental caries in clinical practice? Caries Res. 2004 May-Jun;38(3):294-304. doi: 10.1159/000077769. PMID 15153703
- [Background] Bratthall D. Introducing the Significant Caries Index together with a proposal for a new global oral health goal for 12-year-olds. Int Dent J. 2000 Dec;50(6):378-84. doi: 10.1111/j.1875-595x.2000.tb00572.x. PMID 11197197
- [Background] Ostberg AL. Adolescents' views of oral health education. A qualitative study. Acta Odontol Scand. 2005 Oct;63(5):300-7. doi: 10.1080/00016350510020061. PMID 16419436
- [Background] Grindefjord M, Dahllof G, Nilsson B, Modeer T. Prediction of dental caries development in 1-year-old children. Caries Res. 1995;29(5):343-8. doi: 10.1159/000262090. PMID 8521434
- [Background] Andre Kramer AC, Petzold M, Hakeberg M, Ostberg AL. Multiple Socioeconomic Factors and Dental Caries in Swedish Children and Adolescents. Caries Res. 2018;52(1-2):42-50. doi: 10.1159/000481411. Epub 2017 Dec 14. PMID 29237152
- [Background] Sundgot-Borgen J, Torstveit MK. Prevalence of eating disorders in elite athletes is higher than in the general population. Clin J Sport Med. 2004 Jan;14(1):25-32. doi: 10.1097/00042752-200401000-00005. PMID 14712163
- [Background] Johansson AK, Norring C, Unell L, Johansson A. Diet and behavioral habits related to oral health in eating disorder patients: a matched case-control study. J Eat Disord. 2020 Feb 27;8:7. doi: 10.1186/s40337-020-0281-z. eCollection 2020. PMID 32128206
- [Background] 30. Nilsen H. Alle tannleger må være forberedt på pasienter som misbruker stoff. 2000;110
- [Background] Fagerstad A, Windahl J, Arnrup K. Understanding avoidance and non-attendance among adolescents in dental care - an integrative review. Community Dent Health. 2016 Sep;33(3):195-207. doi: 10.1922/CDH_3829Fagerstad13. PMID 28509515
- [Background] Alm A, Fahraeus C, Wendt LK, Koch G, Andersson-Gare B, Birkhed D. Body adiposity status in teenagers and snacking habits in early childhood in relation to approximal caries at 15 years of age. Int J Paediatr Dent. 2008 May;18(3):189-96. doi: 10.1111/j.1365-263X.2007.00906.x. Epub 2008 Mar 6. PMID 18328046
- [Background] Bradbury KM, Turel O, Morrison KM. Electronic device use and beverage related sugar and caffeine intake in US adolescents. PLoS One. 2019 Oct 22;14(10):e0223912. doi: 10.1371/journal.pone.0223912. eCollection 2019. PMID 31639162
- [Background] Wigen TI, Wang NJ. Characteristics of teenagers who use dental floss. Community Dent Health. 2021 Feb 25;38(1):10-14. doi: 10.1922/CDH_00006Wigen05. PMID 32407009
- [Background] Vaktskjold A. Frequency of tooth brushing and associated factors among adolescents in western Norway. Norsk Epidemiologi. 2019;28:97-103
- [Background] Ericsson JS, Wennstrom JL, Lindgren B, Petzold M, Ostberg AL, Abrahamsson KH. Health investment behaviours and oral/gingival health condition, a cross-sectional study among Swedish 19-year olds. Acta Odontol Scand. 2016;74(4):265-71. doi: 10.3109/00016357.2015.1112424. Epub 2015 Nov 24. PMID 26599291
- [Background] Ericsson JS, Ostberg AL, Wennstrom JL, Abrahamsson KH. Oral health-related perceptions, attitudes, and behavior in relation to oral hygiene conditions in an adolescent population. Eur J Oral Sci. 2012 Aug;120(4):335-41. doi: 10.1111/j.1600-0722.2012.00970.x. Epub 2012 Jun 25. PMID 22813224
- [Background] Skaret E, Raadal M, Kvale G, Berg E. Factors related to missed and cancelled dental appointments among adolescents in Norway. Eur J Oral Sci. 2000 Jun;108(3):175-83. doi: 10.1034/j.1600-0722.2000.108003175.x. PMID 10872986
- [Background] Klingberg G. Dental fear and behavior management problems in children. A study of measurement, prevalence, concomitant factors, and clinical effects. Swed Dent J Suppl. 1995;103:1-78. PMID 7740439
- [Background] Ostberg AL, Ericsson JS, Wennstrom JL, Abrahamsson KH. Socio-economic and lifestyle factors in relation to priority of dental care in a Swedish adolescent population. Swed Dent J. 2010;34(2):87-94. PMID 20701217
- [Background] Wang NJ, Aspelund GO. Children who break dental appointments. Eur Arch Paediatr Dent. 2009 Jan;10(1):11-4. doi: 10.1007/BF03262660. PMID 19254520
- [Background] Holmen TL, Bratberg G, Krokstad S, Langhammer A, Hveem K, Midthjell K, Heggland J, Holmen J. Cohort profile of the Young-HUNT Study, Norway: a population-based study of adolescents. Int J Epidemiol. 2014 Apr;43(2):536-44. doi: 10.1093/ije/dys232. Epub 2013 Feb 4. PMID 23382364
- [Derived] Hovik H, Jensen KHM, Borsting T, Eftedal RK, Dahllof G, Hafell B, Fagerhaug TN, Lassemo E, Hoiseth M, Sen A, Skeie MS. Individual caries increments during adolescence in seven Norwegian cohorts born 1996-2002. BMC Oral Health. 2025 Jun 3;25(1):901. doi: 10.1186/s12903-025-06136-6. PMID 40462067
- See also: Statistics — https://www.ssb.no/statbank/table/11985/
- See also: Mental health report — https://www.fhi.no/globalassets/dokumenterfiler/rapporter/2018/psykisk_helse_i_norge2018.pdf